CLINICAL TRIAL: NCT03004326
Title: Clinical Transcriptomics in Systemic Vasculitis (CUTIS)
Acronym: CUTIS
Status: Recruiting | Type: Observational
Sponsor: Peter Merkel (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH); Office of Rare Diseases Research (ORDR) (Unknown)
Responsible Party: Sponsor-Investigator, Peter Merkel, Chief, Division of Rheumatology Professor of Medicine and Epidemiology, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Other Study IDs: VCRC5563; U54AR057319 (NIH)
Record Dates: First submitted 2016-12-20; First posted 2016-12-28 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Cryoglobulinemic Vasculitis (CV); Drug-induced Vasculitis; Eosinophilic Granulomatosis With Polyangiitis (EGPA); IgA Vasculitis; Isolated Cutaneous Vasculitis; Granulomatosis With Polyangiitis (GPA); Microscopic Polyangiitis (MPA); Polyarteritis Nodosa (PAN); Urticarial Vasculitis; Vasculitis
Keywords: DIV; CSS; EGPA; HSP; GPA; MPA; PAN; Wegeners
MeSH Terms: conditions — Cryoglobulinemia, Familial Mixed; Churg-Strauss Syndrome; IgA Vasculitis; Granulomatosis with Polyangiitis; Microscopic Polyangiitis; Polyarteritis Nodosa; Vasculitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected solely for research purposes. The reason we are performing these laboratory-based research studies is to help us better understand whether abnormalities detected in a subjects skin biopsy can also be detected in their blood.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Multi-center observational study to evaluate the histopathology and transcriptome of cutaneous lesions in patients with several different types of vasculitis.

DETAILED DESCRIPTION:
This study employs a multi-center approach to evaluate cutaneous vasculitis across several forms of idiopathic vasculitis. Patients with cutaneous manifestations of vasculitis will be evaluated by teams of primary vasculitis care providers and Dermatologists in order to facilitate optimal selection of patients and sampling of lesions.

A punch skin biopsy at a site of active vasculitis will be the source of material for histopathologic and transcriptomic evaluation. The histopathology of cutaneous vasculitis will be characterized using a standardized approach.

ELIGIBILITY:
Inclusion Criteria:

* Have a cutaneous lesion (purpuric macules, palpable purpura, retiform purpura, nodules, ulcers, or urticarial) believed to be related to active vasculitis
* Have a suspected or confirmed diagnosis of:

  * Cryoglobulinemic vasculitis (CV)
  * Drug-induced vasculitis
  * Eosinophilic granulomatosis with polyangiitis (EGPA)
  * IgA vasculitis
  * Isolated cutaneous vasculitis
  * Granulomatosis with polyangiitis (GPA)
  * Microscopic polyangiitis (MPA)
  * Polyarteritis nodosa (PAN)
  * Urticarial vasculitis
* Be willing and able to provide written informed consent (or assent for those under

Exclusion Criteria:

* You are less than five years old
* Considered not to be a candidate for a biopsy or have a higher risk of developing an infection, bleeding, etc., from the biopsy, or a doctor believes that the risks for you participating in this study do not outweigh the potential benefit of learning information from your biopsy
* You have a neutrophil count (type of white blood cell) less than 1500/mm3, platelet count less than 50,000/mm3, or a hemoglobin less than 7 g/dL
* You have an uncontrolled disease that could prevent you from completing the study procedures
* You have an active infection at or near the potential biopsy site, have poor circulation, or have bony prominence or other structure that would increase your risk of complications if you participated in this study
* You are pregnant or nursing
* You are not able to provide informed consent

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: About 56 people with vasculitis will take part in this study at approximately 20 medical centers across North America. Patients with CV, DiV, EGPA, IgA vasculitis, GPA, MPA, PAN, isolated cutaneous vasculitis and urticarial vasculitis will potentially be enrolled into this study.
  The protocol will be conducted at the major vasculitis centers in the United States and Canada participating in selected VCRC studies. Skin biopsy specimens collected as standard of care for these diseases will be retrieved and used in research.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of clinical data and linked biopsy specimens | 1 year
  Describe cutaneous vasculitis across several different forms of systemic vasculitis using histopathology.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Micheletti, MD, Principal Investigator — University of Pennsylvania; Peter Grayson, MD, MSc, Principal Investigator — The National Institute of Arthritis and Musculoskeletal and Skin Diseases
Locations (10):
- United States (8):
  - University of California, Los Angeles, Los Angeles, California
  - Boston University School of Medicine, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
- Canada (2):
  - St. Joseph's Healthcare, Hamilton, Ontario
  - University of Toronto Mount Sinai Hospital, Toronto, Ontario

REFERENCES:
- See also: Related Info — http://www.rarediseasesnetwork.org/vcrc